CLINICAL TRIAL: NCT04501120
Title: A Phase Ib Study of the Safety, Pharmacokinetic of Lisaftoclax (APG-2575) Single Agent and in Combination With Homoharringtonine or Azacitidine in Patients With Relapsed/Refractory AML
Brief Title: Study of Lisaftoclax (APG-2575) Single Agent and Combination With Therapy in Patients Relapsed/Refractory AML
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Collaborators: Suzhou Yasheng Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APG2575AC101
Record Dates: First submitted 2020-08-03; First posted 2020-08-06 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Relapsed/Refractory Acute Myeloid Leukaemia; Myeloid Malignancy
Keywords: Acute Myeloid Leukaemia (AML); Bcl-2 Inhibitor; Myeloid Malignancy; Lisaftoclax (APG-2575)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Lisaftoclax; Azacitidine; olverembatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Lisaftoclax (APG-2575) single agent (Experimental): Lisaftoclax (APG-2575) orally once daily starting from 200mg and will be increased in subsequent cohorts to 400mg, 600mg, 800mg, to determine the MTD/RP2D.
  Interventions: Drug: Lisaftoclax (APG-2575)
- Lisaftoclax (APG-2575)+reduced-dose HHT (Experimental): Lisaftoclax (APG-2575) MTD/RP2D-1 and MTD/RP2D combines with reduced-dose HHT in R/R AML, MPAL, BPDCN, CMML.
  Interventions: Drug: Lisaftoclax (APG-2575); Drug: Reduced-dose HHT
- Lisaftoclax (APG-2575)+ standard-dose HHT (Experimental): Lisaftoclax (APG-2575) MTD/RP2D-1 and MTD/RP2D combines with standard-dose HHT in R/R AML, MPAL, BPDCN, CMML.
  Interventions: Drug: Lisaftoclax (APG-2575); Drug: standard-dose HHT
- Lisaftoclax (APG-2575)+ AZA (Experimental): Lisaftoclax (APG-2575) MTD/RP2D-1 and MTD/RP2D combines with AZA in R/R AML, MPAL, BPDCN, CMML.
  Interventions: Drug: Lisaftoclax (APG-2575); Drug: Azacitidine
- Lisaftoclax (APG-2575)+ AZA(HR-MDS.) (Experimental): Lisaftoclax (APG-2575) MTD/RP2D-1 and MTD/RP2D combines with AZA in HR-MDS.
  Interventions: Drug: Azacitidine; Drug: Lisaftoclax (APG-2575)
- Lisaftoclax (APG-2575)+ AZA(Naïve AML.) (Experimental): Lisaftoclax (APG-2575) MTD/RP2D-1 and MTD/RP2D combines with AZA in treatment naïve AML.
  Interventions: Drug: Lisaftoclax (APG-2575); Drug: Azacitidine
- Lisaftoclax (APG-2575)+AZA+Olverembatinib (Experimental): Lisaftoclax (APG-2575) combines with AZA and Olverembatinib in R/R AML.
  Interventions: Drug: Azacitidine; Drug: Lisaftoclax (APG-2575); Drug: olverembatinib
- Lisaftoclax (APG-2575)+HHT+Olverembatinib (Experimental): Lisaftoclax (APG-2575) combines with HHT and Olverembatinib in R/R AML.
  Interventions: Drug: standard-dose HHT; Drug: Lisaftoclax (APG-2575); Drug: olverembatinib

INTERVENTIONS:
Drug: Lisaftoclax (APG-2575) — Lisaftoclax (APG-2575) orally once daily, every 28 days as a cycle.
  Arms: Lisaftoclax (APG-2575) single agent; Lisaftoclax (APG-2575)+ AZA; Lisaftoclax (APG-2575)+ AZA(Naïve AML.); Lisaftoclax (APG-2575)+ standard-dose HHT; Lisaftoclax (APG-2575)+reduced-dose HHT
Drug: Reduced-dose HHT — 1mg IV QD on Days 1-14 (28-day cycle).
  Arms: Lisaftoclax (APG-2575)+reduced-dose HHT
Drug: standard-dose HHT — 2mg/m^2 IV QD on Days 1-7 (28-day cycle).
  Arms: Lisaftoclax (APG-2575)+ standard-dose HHT; Lisaftoclax (APG-2575)+HHT+Olverembatinib
Drug: Azacitidine — 75 mg/m^2 SC or Iv gtt QD on Days 1- 7 (28-day cycle).
  Arms: Lisaftoclax (APG-2575)+ AZA; Lisaftoclax (APG-2575)+ AZA(HR-MDS.); Lisaftoclax (APG-2575)+ AZA(Naïve AML.); Lisaftoclax (APG-2575)+AZA+Olverembatinib
Drug: Lisaftoclax (APG-2575) — Lisaftoclax (APG-2575) orally once daily for 14 days, every 28 days as a cycle.
  Arms: Lisaftoclax (APG-2575)+ AZA(HR-MDS.); Lisaftoclax (APG-2575)+AZA+Olverembatinib; Lisaftoclax (APG-2575)+HHT+Olverembatinib
Drug: olverembatinib — orally, with meals, QOD, every 28 days as a cycle.
  Arms: Lisaftoclax (APG-2575)+AZA+Olverembatinib; Lisaftoclax (APG-2575)+HHT+Olverembatinib

SUMMARY:
The purpose of this study is to assess the safety, pharmacokinetic profile of Lisaftoclax (APG-2575) single agent and in combination with HHT/AZA in patients with relapsed/refractory AML and related myeloid malignancies.

DETAILED DESCRIPTION:
This is an open-label, multi-center Phase Ib study of safety, PK of Lisaftoclax (APG-2575) as single agent or in combination with HHT or AZA in relapsed/refractory AML and related myeloid malignancies patients.

This study consists of three stages: The first stage is the Lisaftoclax (APG-2575) single agent dose-escalation study. The second stage is the Lisaftoclax (APG-2575) combined with HHT/AZA dose-escalation study. The third stage is the MTD/RP2D expansion cohort study of the combination regimen.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet each of the following inclusion criteria are eligible to participate in this study:

1. In accordance with the World Health Organization (WHO) 2016 diagnostic criteria for relapsed or refractory acute myeloid leukemia (AML), Mixed phenotype acute leukemia(MPAL), Chronic myelomonocytic leukemia (CMML), Higher-risk myelodysplastic syndrome (HR-MDS) , Blastic plasmacytoid dendritic cell neoplasm (BPDCN) and naïve AML ineligible for treatment with a standard chemotherapy due to age or comorbidities.
2. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS): 0 -2 (0 to 3 for participants >= 60 to 74 years of age who are evaluated as ineligible for treatment with standard chemotherapy).
3. Subjects can accept oral administration of Lisaftoclax (APG-2575).
4. Life expectancy ≥ 3 months.
5. Adequate renal and liver function.
6. Males, female patients of childbearing potential (postmenopausal women who must have been menopausal for at least 12 months to be considered infertile) and their partners voluntarily take contraception which the investigator considers effective during treatment and at least three months after the last dose of study drug.
7. Ability to understand and willingness to sign a written informed consent form (the consent form must be signed by the patient prior to any study-specific procedures).
8. Willingness and ability to comply with study procedures and follow-up examination.

Exclusion Criteria:

Patients who meet any of the following exclusion criteria are not to be enrolled in this study:

1. Patients diagnosed with acute promyelocytic leukemia or t(9;22)(q34.1;q11.2); BCR-ABL1 positive AML patients.
2. The persistent toxicities caused by previous chemotherapy or radiotherapy has not been restored to lower than grade 2 by CTCAE 5.0 (except for alopecia).
3. Known leukemia infiltration of the central nervous system.
4. Symptomatic active fungal, bacterial and/or viral infections.
5. Prior history of allogeneic hematopoietic stem cell transplantation or adoptive cell immunotherapy, autologous hematopoietic stem cell transplantation within 12 months.
6. Within 14 days before the first dose of study drug, received chemotherapy (hydroxyurea is permitted more than 24 hours before the first dose of study drug), radiotherapy, surgery, immunotherapy, targeted therapy, biological therapy or any investigational treatment.
7. Within 7 days before the first dose of study drug, received a strong and/or moderate CYP3A inducer and/or Inhibitor.
8. At the discretion of the investigator, gastrointestinal diseases that affect the absorption of Lisaftoclax (APG-2575).
9. Any other condition or circumstance, at the discretion of the investigator, that patients would be unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Estimated)
Dates: Start 2020-09-28 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | 28 days
  DLT will be graded according to NCI CTCAE Version 5.0. DLT will be defined as clinically significant drug-related adverse events during cycle one.
Maximum Tolerated Dose (MTD)/Recommended Phase 2 Dose(RP2D) | 28 days
  MTD/RP2D will be determined based on DLTs observed during cycle one.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | 28 days
  Cmax of Lisaftoclax (APG-2575) will be assessed in the patients in single agent or combo study.
Area under the plasma concentration versus time curve (AUC) | 28 days
  AUC of Lisaftoclax (APG-2575) will be assessed in the patients in single agent or combo study.
Objective Response Rate (ORR) | Up to 6 cycles (each cycle is 28 days).
  ORR is defined by CR+ CRi + PR(according to IWG AML(2003)).Response will be evaluated on cycle 1 and every even cycles till completing 6 cycles treatment or end of treatment.
progression free survival (PFS) | Up to 2 years.
  From date of treatment start until the date of progression or the date of death due to any cause.
duration of response (DOR) | Up to 2 years.
  From date of response until the date of progression.
overall survival (OS) | Up to 2 years.
  From date of treatment start until the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Yifan Zhai, M.D., Ph.D., Study Director — Suzhou Yasheng Pharmaceutical Co., Ltd.; Jie Jin, M.D., Principal Investigator — the First Affiliated Hospital, College of Medicine
Locations (12):
- China (12):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guandong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Henan Tumor Hospital, Zhengzhou, Henan
  - Union Hospital medical college Huazhong University of Science and Technology, Wuhan, Hubei
  - Zhongnan Hospital of Hunan university, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The First affiliated hospital of Soochow University, Suzhou, Jiangsu
  - Shanghai The Sixth People' s Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - the First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang